CLINICAL TRIAL: NCT03034642
Title: Modulation of Steroid Immunosuppression by Alveolar Efferocytosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey Curtis, Staff Physician, VA Ann Arbor Healthcare System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VAAAHS Curtis 0038; I01CX000911 (NIH)
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Pneumonia, Bacterial
Keywords: Apoptosis; Bronchoscopy; Human; Mice, inbred strains; Macrophages, Alveolar; MicroRNAs; Streptococcus pneumoniae; Fluticasone
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia, Bacterial | interventions — Bronchoscopy

STUDY DESIGN:
Intervention Model Description: This study will analyze both healthy subjects (never-smokers and current- or ex-smokers) in one arm, and also subjects with COPD (current- or ex-smokers).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (Experimental): Procedure/Surgery: Bronchoscopy with bilateral bronchoalveolar lavages.
  Drugs: No test substances, only moderate conscious sedation using standard medications.
  Devices: No test devices.
  Interventions: Procedure: Bronchoscopy with bilateral bronchoalveolar lavages
- COPD participants (Experimental): Procedure/Surgery: Bronchoscopy with bilateral bronchoalveolar lavages.
  Drugs: No test substances, only moderate conscious sedation using standard medications.
  Devices: No test devices.
  Interventions: Procedure: Bronchoscopy with bilateral bronchoalveolar lavages

INTERVENTIONS:
Procedure: Bronchoscopy with bilateral bronchoalveolar lavages — Bronchoscopy with bilateral bronchoalveolar lavages

SUMMARY:
The long-term goals of this study are (a) to understand the biological underpinnings for the increased incidence of community-acquired pneumonia in patients with chronic obstructive pulmonary disease (COPD) who are treated with inhaled corticosteroids; and (b) to develop novel therapies to treated this problem using over-expression of micro-RNAs (miRNAs).

DETAILED DESCRIPTION:
Treating chronic obstructive pulmonary disease (COPD) patients with inhaled glucocorticosteroids has been convincingly shown to increase their risk of pneumonia, but the responsible mechanisms are undefined. Work from this laboratory suggests a possible mechanism, related to the increased numbers of cells dying by apoptosis in the lungs in COPD, especially in emphysema. Uptake of apoptotic cells ("efferocytosis") suppresses the ability of alveolar macrophages (AM) to fight infections. By markedly increasing AM efferocytosis, glucocorticoids plus apoptotic cells cause greater immune defects than either stimulus alone. These defects include reductions in killing of Streptococcus pneumoniae by human AM and murine AM in vitro, and in clearance of viable pneumococci from lungs of mice. This effect is called glucocorticoid augmented efferocytosis (GCAE). MicroRNAs (miRNAs) are 19-25 nucleotide-long non-coding RNAs that coordinately target large numbers of genes and reduce their protein products. Preliminary data imply that defective AM function is caused by down-regulation of specific miRNAs by GCAE (but not by apoptotic cells alone or glucocorticosteroids alone). The long-term goal of this project is to develop novel inhalational treatments based on transient over-expression of these specifically decreased miRNAs, to reverse defective AM immune function when COPD patients taking inhaled glucocorticoids present with community-acquired pneumonia. This project will use both ex vivo investigation of AM from human volunteers (never-smokers; smokers with normal spirometry; and COPD subjects who are current or former smokers), and an established murine model of pneumococcal pneumonia. Its immediate goals are to: (a) confirm that GCAE increases pneumococcal pneumonia risk and severity, and in the process, validate a murine model for testing strategies to reverse those defects; (b) define GCAE-induced AM defects functionally and by whole-transcriptome analysis, identifying genes and miRNAs uniquely regulated by the GCAE x pneumococcus interaction; (c) validate and optimize miRNA-over-expression to reverse the adverse effects of GCAE on AM defensive functions. Successful completion of this project could lead to more precisely personalized therapies and better outcomes in COPD, currently the third leading cause of death in the USA

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for healthy subjects without COPD:
* Age 18-80 years, inclusive
* Males or females
* Never smoker (< 100 cigarettes in lifetime)

  * OR
* Current smoker (>10 pack-years) with normal spirometry
* Able to perform satisfactory spirometry
* Abe to give informed consent
* Able to complete questionnaires
* Inclusion Criteria for COPD subjects:
* Age 18-80 years, inclusive
* Males or females
* Current smoker

  * (>10 pack-years) & (≥1/2 pack/day)

    * OR
* Former smoker

  * (>10 pack-years) & (>6 months of non-smoking)
* Diagnosis of COPD by ATS/ERS1 criteria
* Able to perform satisfactory spirometry
* Able to give informed consent
* Able to complete questionnaires
* 1 ATS/ERS, American Thoracic Society/European Respiratory Society.

Exclusion Criteria:

* Exclusion Criteria for healthy subjects without COPD:
* Unstable cardiovascular disease, including uncontrolled hypertension, CHF, angina
* Significant renal (creatinine >2.5) or hepatic dysfunction (Childs B or C)
* Mental incompetence/active psychiatric illness
* Prednisone or other immunosuppressive medications
* Participation in another interventional experimental protocol within 6 weeks
* Pregnancy
* Use of antibiotics for any reason within 42 days
* Judged to be unsuitable for bronchoscopy by PI
* Resting SaO2<93%
* FEV1 < 70% predicted
* Respiratory infections within 42 days regardless of antibiotic use
* Diagnosed COPD or Asthma
* Use of inhaled corticosteroids
* Active pulmonary tuberculosis or other serious chronic respiratory infection
* Diffuse panbronchiolitis or Cystic fibrosis
* Clinically significant bronchiectasis
* History of thoracic radiation therapy for any cause
* Other inflammatory or fibrotic lung disease
* Exclusion Criteria for COPD subjects:
* Unstable cardiovascular disease, including uncontrolled hypertension, CHF, angina
* Significant renal (creatinine >2.5) or hepatic dysfunction (Childs B or C)
* Mental incompetence/active psychiatric illness
* Prednisone or other immunosuppressive medications
* Participation in another interventional experimental protocol within 6 weeks
* Pregnancy
* Use of antibiotics for any reason within 42 days
* Judged to be unsuitable for bronchoscopy by PI
* Resting daytime SaO2<90% while breathing room air
* FEV1 < 50% predicted
* Respiratory infections within 42 days regardless of antibiotic use
* Use of inhaled corticosteroids
* Active pulmonary tuberculosis or other serious chronic respiratory infection
* Diffuse panbronchiolitis or Cystic fibrosis
* Clinically significant bronchiectasis
* History of thoracic radiation therapy for any cause
* Other inflammatory or fibrotic lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Bactericidal activity of human alveolar macrophage against S. pneumoniae in vitro | 24 hours
  Alveolar macrophages from volunteers will be be assayed for their ability to kill pneumococci in vitro following treatment with glucocorticoids, apoptotic cells or both. Participation of the subjects ends after bronchoscopy, and no clinical outcomes will be measured.

SECONDARY OUTCOMES:
Mechanisms of human alveolar macrophage killing of S. pneumoniae in vitro | 24 hours
  These same macrophages will also be assayed for production of mRNA and regulatory microRNAs (by RNA sequencing and quantitative real-time PCR and for cytokine and chemokine production.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Curtis, M.D., Principal Investigator — University of Michigan
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCubbrey AL, Sonstein J, Ames TM, Freeman CM, Curtis JL. Glucocorticoids relieve collectin-driven suppression of apoptotic cell uptake in murine alveolar macrophages through downregulation of SIRPalpha. J Immunol. 2012 Jul 1;189(1):112-9. doi: 10.4049/jimmunol.1200984. Epub 2012 May 21. PMID 22615206
- [Background] Freeman CM, Martinez CH, Todt JC, Martinez FJ, Han MK, Thompson DL, McCloskey L, Curtis JL. Acute exacerbations of chronic obstructive pulmonary disease are associated with decreased CD4+ & CD8+ T cells and increased growth & differentiation factor-15 (GDF-15) in peripheral blood. Respir Res. 2015 Aug 5;16(1):94. doi: 10.1186/s12931-015-0251-1. PMID 26243260
- [Background] Adar SD, Huffnagle GB, Curtis JL. The respiratory microbiome: an underappreciated player in the human response to inhaled pollutants? Ann Epidemiol. 2016 May;26(5):355-9. doi: 10.1016/j.annepidem.2016.03.010. Epub 2016 Apr 7. PMID 27161078
- [Background] Huang YJ, Erb-Downward JR, Dickson RP, Curtis JL, Huffnagle GB, Han MK. Understanding the role of the microbiome in chronic obstructive pulmonary disease: principles, challenges, and future directions. Transl Res. 2017 Jan;179:71-83. doi: 10.1016/j.trsl.2016.06.007. Epub 2016 Jun 23. PMID 27392936
- [Background] Freeman CM, Curtis JL. Lung Dendritic Cells: Shaping Immune Responses throughout Chronic Obstructive Pulmonary Disease Progression. Am J Respir Cell Mol Biol. 2017 Feb;56(2):152-159. doi: 10.1165/rcmb.2016-0272TR. PMID 27767327
- [Background] Verhamme FM, Freeman CM, Brusselle GG, Bracke KR, Curtis JL. GDF-15 in Pulmonary and Critical Care Medicine. Am J Respir Cell Mol Biol. 2019 Jun;60(6):621-628. doi: 10.1165/rcmb.2018-0379TR. PMID 30633545
- [Background] Freeman CM, Curtis JL. It's Complicated: Lung Dendritic Cells in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2020 Aug 15;202(4):479-481. doi: 10.1164/rccm.202004-0899ED. No abstract available. PMID 32286855
- [Background] Polverino F, Curtis JL. The ABCs of Granulomatous Lung Diseases: Age-associated B Cells. Am J Respir Crit Care Med. 2020 Oct 1;202(7):922-924. doi: 10.1164/rccm.202006-2261ED. No abstract available. PMID 32603192
- [Background] He Y, Wang H, Zheng J, Beiting DP, Masci AM, Yu H, Liu K, Wu J, Curtis JL, Smith B, Alekseyenko AV, Obeid JS. OHMI: the ontology of host-microbiome interactions. J Biomed Semantics. 2019 Dec 30;10(1):25. doi: 10.1186/s13326-019-0217-1. PMID 31888755
- [Background] Tighe RM, Redente EF, Yu YR, Herold S, Sperling AI, Curtis JL, Duggan R, Swaminathan S, Nakano H, Zacharias WJ, Janssen WJ, Freeman CM, Brinkman RR, Singer BD, Jakubzick CV, Misharin AV. Improving the Quality and Reproducibility of Flow Cytometry in the Lung. An Official American Thoracic Society Workshop Report. Am J Respir Cell Mol Biol. 2019 Aug;61(2):150-161. doi: 10.1165/rcmb.2019-0191ST. PMID 31368812
- [Background] Curtis JL. B Cells Caught in the Act: Class Switching to IgA in Lung Lymphoid Follicles in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2019 Mar 1;199(5):548-550. doi: 10.1164/rccm.201810-1907ED. No abstract available. PMID 30352169
- [Result] Stolberg VR, McCubbrey AL, Freeman CM, Brown JP, Crudgington SW, Taitano SH, Saxton BL, Mancuso P, Curtis JL. Glucocorticoid-Augmented Efferocytosis Inhibits Pulmonary Pneumococcal Clearance in Mice by Reducing Alveolar Macrophage Bactericidal Function. J Immunol. 2015 Jul 1;195(1):174-84. doi: 10.4049/jimmunol.1402217. Epub 2015 May 18. PMID 25987742
- [Result] McCubbrey AL, Nelson JD, Stolberg VR, Blakely PK, McCloskey L, Janssen WJ, Freeman CM, Curtis JL. MicroRNA-34a Negatively Regulates Efferocytosis by Tissue Macrophages in Part via SIRT1. J Immunol. 2016 Feb 1;196(3):1366-75. doi: 10.4049/jimmunol.1401838. Epub 2015 Dec 30. PMID 26718338
- [Result] Dickson RP, Erb-Downward JR, Freeman CM, McCloskey L, Beck JM, Huffnagle GB, Curtis JL. Spatial Variation in the Healthy Human Lung Microbiome and the Adapted Island Model of Lung Biogeography. Ann Am Thorac Soc. 2015 Jun;12(6):821-30. doi: 10.1513/AnnalsATS.201501-029OC. PMID 25803243
- [Result] Dickson RP, Erb-Downward JR, Freeman CM, McCloskey L, Falkowski NR, Huffnagle GB, Curtis JL. Bacterial Topography of the Healthy Human Lower Respiratory Tract. mBio. 2017 Feb 14;8(1):e02287-16. doi: 10.1128/mBio.02287-16. PMID 28196961
- [Result] Dickson RP, Erb-Downward JR, Prescott HC, Martinez FJ, Curtis JL, Lama VN, Huffnagle GB. Intraalveolar Catecholamines and the Human Lung Microbiome. Am J Respir Crit Care Med. 2015 Jul 15;192(2):257-9. doi: 10.1164/rccm.201502-0326LE. No abstract available. PMID 26177175
- [Result] Mancuso P, Curtis JL, Freeman CM, Peters-Golden M, Weinberg JB, Myers MG Jr. Ablation of the leptin receptor in myeloid cells impairs pulmonary clearance of Streptococcus pneumoniae and alveolar macrophage bactericidal function. Am J Physiol Lung Cell Mol Physiol. 2018 Jul 1;315(1):L78-L86. doi: 10.1152/ajplung.00447.2017. Epub 2018 Mar 22. PMID 29565180
- [Result] Finch DK, Stolberg VR, Ferguson J, Alikaj H, Kady MR, Richmond BW, Polosukhin VV, Blackwell TS, McCloskey L, Curtis JL, Freeman CM. Lung Dendritic Cells Drive Natural Killer Cytotoxicity in Chronic Obstructive Pulmonary Disease via IL-15Ralpha. Am J Respir Crit Care Med. 2018 Nov 1;198(9):1140-1150. doi: 10.1164/rccm.201712-2513OC. PMID 29676596
- [Result] Erb-Downward JR, Falkowski NR, D'Souza JC, McCloskey LM, McDonald RA, Brown CA, Shedden K, Dickson RP, Freeman CM, Stringer KA, Foxman B, Huffnagle GB, Curtis JL, Adar SD. Critical Relevance of Stochastic Effects on Low-Bacterial-Biomass 16S rRNA Gene Analysis. mBio. 2020 Jun 9;11(3):e00258-20. doi: 10.1128/mBio.00258-20. PMID 32518181
- [Result] Yue M, Kim JH, Evans CR, Kachman M, Erb-Downward JR, D'Souza J, Foxman B, Adar SD, Curtis JL, Stringer KA. Measurement of Short-Chain Fatty Acids in Respiratory Samples: Keep Your Assay above the Water Line. Am J Respir Crit Care Med. 2020 Aug 15;202(4):610-612. doi: 10.1164/rccm.201909-1840LE. No abstract available. PMID 32343599